CLINICAL TRIAL: NCT04830683
Title: Endothelial Dysfunction and Oxidative Stress in ICU and Non-ICU Covid-19 Patients With Hypoxemic Respiratory Failure
Brief Title: Endothelial Dysfunction in Covid-19
Acronym: ENDOCOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/27AVR/247
Record Dates: First submitted 2021-03-26; First posted 2021-04-05 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Covid19; Hypoxemic Respiratory Failure
Keywords: Endothelial Dysfunction; Covid19
MeSH Terms: conditions — COVID-19; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Biospecimen Retention: Samples Without DNA — serum and plasma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ICU Covid-19 patients: Covid-19 patients admitted for refractory respiratory failure despite conventional oxygen therapy requiring Intensive Care Unit (ICU) admission and oxygenation through either High Flow Nasal Cannula (HFNC) therapy or endotracheal intubation with mechanical ventilation
- non-ICU Covid-19 patients: Covid-19 patients admitted at hospital requiring conventional oxygen or continuous positive airways pressure (cpap)
- matched control subjects: Healthy subjects matched for similar cardiovascular risk factors than ICU Covid-19 patients
- ICU septic shock patients: Septic shock patients corresponded to refractory hypotension in response to an infection, in non Covid-19 patients, requiring ICU hospitalisation for vasopressors to maintain mean arterial pressure (MAP) > 65mm Hg despite adequate volume resuscitation according to the Surviving Sepsis Campaign

SUMMARY:
SARS-CoV-2 targets endothelial cells via the angiotensin-converting enzyme 2 receptor. The specific impact of the resulting endothelial injury is currently unknown but may contribute to the pro-coagulant state classically described during Covid-19 disease and commonly associated with an exacerbated activation of the renin-angiotensin-aldosterone system.

DETAILED DESCRIPTION:
We prospectively compared clinical and biological parameters in ICU- and non-ICU-admitted Covid-19 patients, ICU-admitted patients with septic shock unrelated to Covid-19 and matched control subjects.

Primary hemostasis and coagulation parameters and endothelial biomarkers are measured. Activation of the renin-angiotensin-aldosterone system is monitored through measurements of plasma renin, angiotensin II, aldosterone, and serum soluble angiotensin-converting enzyme 2. Vascular oxidative status is assessed by measuring plasma lipids peroxides. Neutrophilic polymorphonuclear activation is assessed by measuring plasma levels of Triggering receptor expressed on myeloid cells-1. Vascular nitric oxide bioavailability is measured by quantification of the concentration of heme-nitrosylated hemoglobin (HbNO) in venous erythrocytes using Electron Paramagnetic Resonance spectroscopy. Structural abnormalities of vascular endothelial cells were analyzed by Transmission Electron- and Scanning Electron Microscopy.

ELIGIBILITY:
Inclusion Criteria:

* positive result on a reverse-transcriptase-polymerase chain reaction testing performed on nasopharyngeal swab at hospital admission

Exclusion Criteria:

* ICU admission more than five days after admission on a general ward,
* concomitant bacterial infection
* older than 75 years
* cirrhosis

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients for SARS-Cov-2 infection
Sampling Method: Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Vascular oxidative stress in Covid-19 versus septic shock and control patients | ICU or general ward hospital admission
  HbNO (nmol/L) and NOX levels (μM/L), oxidative stress with plasma lipids peroxides (mmol/L) levels and soluble TREM-1 measurements. Blood HbNO levels directly correlate with endothelial function and inversely with major cardiovascular risk factors. The nitrite/nitrate levels (NOx) are the the stable end products of NO metabolism that also suggest NO production. Plasma lipids peroxides reflets the surrounding endovascular oxidative stress. sTREM-1 participates in the sepsis-induced ROS production through activation of NADPH oxidase (NOX)-2 during the respiratory burst of activated polymorphonuclear.

SECONDARY OUTCOMES:
Vascular Renin-angiotensin-aldosterone system measurements in Covid-19 versus septic shock and control patients | ICU or general ward hospital admission
  Renin (pg/mL), Agiotensin II (fmol/mL), Aldosterone (pg/mL) measurements. The RAAS system is a classical activator of vascular NOX2 and ROS production.

CONTACTS AND LOCATIONS:
Overall Officials: VIRGINIE MONTIEL, MD,PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Belgique, Belgium

IPD SHARING:
Plan to Share IPD: No